CLINICAL TRIAL: NCT04671693
Title: Study of Complications Related to Treatments in Adults Aged 18 to 65 Years Old Responding to a First Treatment in Oncology or Onco-hematology and Participating in the PASCA (PArcours de Santé au Cours du CAncer) Post-treatment Program.
Brief Title: A Post-treatment Program to Identify and Manage Complications Related to Oncology or Hematology Treatments in Cancer Survivors.
Acronym: PASCA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Malakoff-Humanis (Unknown); Fondation Apicil (Other); Fédération Leucémie Espoir (Unknown); Biogaran (Unknown); Le défi Anthony (Unknown); Novartis (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PASCA; 2020-A01130-39 (Registry Identifier: IDRCB - French Agency for the Safety of Health Products)
Record Dates: First submitted 2020-12-03; First posted 2020-12-17 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Late Effects; Testicular Germ Cell Tumor Mixed; Non-Metastatic Breast Carcinoma; Soft Tissue Sarcoma, Adult, Stage IIC; Osteosarcoma; Ewing's Sarcoma; Acute Myeloid Leukemia; Hodgkin Disease; Non Hodgkin Lymphoma
Keywords: Late Effects; Survivors; Adults; Screening; Tertiary prevention; Testicular Germ Cell Tumor Mixed; Non-Metastatic Breast Carcinoma; Soft Tissue Sarcoma; Osteosarcoma; Ewing's Sarcoma; Acute Myeloid Leukemia; Hodgkin Disease; Non Hodgkin Lymphoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma; Sarcoma, Ewing; Leukemia, Myeloid, Acute; Hodgkin Disease; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Intervention Model Description: All patients in the study will benefit from the PASCA post-treatment program with 4 visits : at 1 month (T1), 6 month (T2), 24 month (T3) and 60 month (T4) after the end of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PASCA intervention (Experimental)
  Interventions: Other: PASCA intervention

INTERVENTIONS:
Other: PASCA intervention — At each study visit (T1 = 1 month, T2 = 6 months, T3 = 24 months, T4 = 60 months), an exhaustive screening of complications as well as associated sub-clinical abnormalities and risk factors previously identified as such in the literature, will be conducted.
  Management of complications consists of referring the patient to a healthcare professional belonging to the PASCA network based on the test results. Referral is defined by referring to pre-established decision trees. It is made to a specialist physician, a health professional from the paramedical field or the patient's general practitioner who confirms the diagnosis if necessary and initiates the patient's care and follow-up. These patients also receive their usual follow-up in the context of their tumor pathology in oncology and onco-hematology.

SUMMARY:
INTRODUCTION: Approximately 44% of cancer survivors experience a deteriorated quality of life 5 years after diagnosis due to late onset of complications related to cancer treatments. The objective of the study is to evaluate the incidence rates of treatment-related complications, identify sub-clinical abnormalities and risk factors in patients participating in the PASCA post-treatment program.

METHOD: PASCA is a single-center, interventional cohort study of adult patients who received at least chemotherapy and with a complete remission to a testicular germ cell tumor, primary non-metastatic invasive breast carcinoma, high-grade soft tissue sarcoma, osteosarcoma, Ewing's sarcoma, acute myeloid leukemia, Hodgkin's or aggressive non-Hodgkin's lymphoma. Four assessment visits will be scheduled at 1 month (T1), 6 months (T2), 24 months (T3) and 60 months (T4) after completion of treatment. During these visits, 19 complications will be screened and follow-up care will be systematically offered to the health professional concerned by the complication in case of a positive result. The screening will contain the following elements: screening self-questionnaires, quality of life questionnaire, 12 biological parameters, a urinalysis evaluating hematuria, proteinuria, and leukocyturia, a spirometry, an electrocardiogram, 5 tests evaluating physical condition, vital signs and the perimetric measurement between both arms.

DISCUSSION: This systematic screening could highlight a number of complications occurring after cancer treatments. Sub-clinical abnormalities and new risk factors could also be identified. This new organization of care could improve the quality of life of adult cancer survivors.

ELIGIBILITY:
1. males and females aged 18-65 years;
2. Diagnosis and management at CLB for one of the following cancers: Hodgkin's lymphoma, aggressive non-Hodgkin's lymphoma, acute myeloid leukemia and primary non metastatic invasive breast cancer (BC), TGCT, or Sarcoma (Soft Tissue Sarcoma, Osteosarcoma, and Ewing's Sarcoma);
3. receiving first-line intensive chemotherapy;
4. with a complete response status at the end of the last treatment, which may include chemotherapy (excluding maintenance and hormone therapy), radiotherapy or adjuvant surgery, depending on the last scheduled treatment;
5. No contraindications to adapted physical activity (APA) at inclusion;
6. no medical, social, family, or psychological barriers against study participation.

Patients will be excluded if they have a history or coexistence of another primary cancer (except basal cell skin cancer), are participating in another study affecting the primary outcome, are deprived of liberty, or reside outside the Auvergne-Rhône-Alpes region or the Saône-et-Loire department.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2029-01-24 (Estimated); Study Completion 2029-04-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of social precariousness | Month 1
  Diagnosed by a social worker
Change from Baseline return to work issues incidence at 60 months | Month 1, Month 6, Month 24, Month 60
  Diagnosed by a social worker
Change from Baseline cognitive problems incidence at 60 months | Month 1, Month 6, Month 24, Month 60
  Diagnosed by a neurologist
Change from Baseline anxiety crises incidence at 60 months | Month 1, Month 6, Month 24, Month 60
  Diagnosed by a psychologist or psychiatrist
Change from Baseline depressive events incidence at 60 months | Month 1, Month 6, Month 24, Month 60
  Questionnaire "HADS-D" (Hospital Anxiety and Depression scale)
Change from Baseline physical deconditioning incidence at 60 months | Month 1, Month 6, Month 24, Month 60
  A value below the lower limit on at least two of the following physical tests
  * Six-Minute Walk Test (6MWT) (meters)
  * Hand Grip Strength Test (Kg)
  * Five Times Sit to Stand Test (number)
  * Flamingo Test (sec)
Change from Baseline overweight/obesity incidence at 60 months | Month 1, Month 6, Month 24, Month 60
  * BMI
  * Waist circumference
Change from Baseline chronic pain incidence at 60 months | Month 1, Month 6, Month 24, Month 60
  * Duration of pain
  * Questionnaire "DN4" (Douleur Neuropathique en 4 questions)
Change from Baseline dermatological disorders incidence at 60 months | Month 1, Month 6, Month 24, Month 60
  Common Terminology Criteria for Adverse Events (CTCAE) v5
Change from Baseline gastrointestinal disorders incidence at 60 months | Month 1, Month 6, Month 24, Month 60
  Common Terminology Criteria for Adverse Events (CTCAE) v5
Change from Baseline sexual disorders incidence at 60 months | Month 1, Month 6, Month 24, Month 60
  Questionnaire "Sexualité VICAN5"
Change from Baseline hypogonadism incidence at 60 months | Month 1, Month 6, Month 24, Month 60
  Presence of clinical signs as defined by the International Society for Sexual Medicine
  A value below the lower limit on at least one of the following blood assay:
  * level of total testosterone
  * level of bioavailable testosterone
Change from 24 months premature ovarian failure incidence at 60 months | Month 24, Month 60
  * level of Follicle stimulating hormone
  * level of estradiol
Change from Baseline osteoporosis incidence at 60 months | Month 1, Month 6, Month 24, Month 60
  T-score evaluated by osteodensitometry, on the lumbar spine and upper end of the femur
Change from Baseline chronic kidney failure incidence at 60 months | Month 1, Month 6, Month 24, Month 60
  Diagnosed on the basis of 2 blood tests within 3 months using the same technique showing a decrease in GFR to < 60ml/min/1.73m2, estimated from creatinine levels using the CKD-EPI equation (Chronic Kidney Disease EPIdemiology collaboration, Levey, 2009), albuminuria or proteinuria positive, hematuria, leukocyturia > 10/mm3, or morphological abnormality on renal ultrasound.
Change from Baseline heart failure incidence at 60 months | Month 1, Month 6, Month 24, Month 60
  Diagnosed by a cardiologist with an echocardiography performing the Left Ventricular Ejection Fraction (LVEF) estimate
Change from Baseline coronary heart disease incidence at 60 months | Month 1, Month 6, Month 24, Month 60
  Diagnosed by a cardiologist conducting at least an interrogation with clinical examination, an estimation of pre-test probability of coronary artery disease
Change from Baseline respiratory failure incidence at 60 months | Month 1, Month 6, Month 24, Month 60
  * Forced Vital Capacity
  * Forced expiratory volume in 1 second
  * Vital capacity
  * Tiffeneau ratio
  * Peak expiratory flow
  * Total lung capacity
  * Diffusing Capacity Of The Lungs For Carbon Monoxide
Change from Baseline hypothyroidism incidence at 60 months | Month 1, Month 6, Month 24, Month 60
  * level of thyroid-stimulating hormone
  * level of total thyroxine

SECONDARY OUTCOMES:
Evaluate the PASCA program: referrals made through the network | Month 6, Month 24, Month 60
  Number of referrals made through the network (attending physicians, specialist physicians, supportive care services or other health professionals)
Evaluate the PASCA program: time between patient referral and completion of the first consultation | Month 6, Month 24, Month 60
  Average time (days) between patient referral and completion of the first consultation
Evaluate the PASCA program: patients description | Month 1, Month 6, Month 24, Month 60
  * Comorbidities at diagnosis
  * Tumor classification
  * types and doses of each cancer treatments
  * ratio of the number of patients included / number of eligible patients
Evaluation of the patient adherence | Month 1, Month 6, Month 24, Month 60
  Ratio of the number of prescriptions issued for referral consultations /number of referral consultations actually attended by the patient
Description of the PASCA network : characteristics of health professionals sensitive to the post-treatment issues. | Month 6, Month 24, Month 60
  * number of health professionals affiliated with the network
  * type of health professionals affiliated with the network
  * distribution over the Auvergne-Rhône-Alpes region according to medical speciality and department
Identification of risk factors associated with complications occurring during follow-up. | Month 1, Month 6, Month 24, Month 60
  Measurement of the association between suspected risk factors and the occurrence of a type of complication, during the duration of follow-up.
Description of the Global Longitudinal Strain | Month 6, Month 24, Month 60
  Evolution of the Global Longitudinal Strain in absolute value, relative to a later value
Description of the troponin I level | Month 6, Month 24, Month 60
  Evolution of the troponin I level relative to a later value
Description of the Glomerular Filtration Rate | Month 6, Month 24, Month 60
  Evolution of the Glomerular Filtration Rate estimated by the CKD-EPI equation relative to a later value
Description of spirometry values | Month 6, Month 24, Month 60
  Evolution of spirometry values relative to later values :
  * Forced Vital Capacity
  * Forced expiratory volume in 1 second
  * Vital capacity
  * Tiffeneau ratio
  * Peak expiratory flow
Incidence of diabetes mellitus | Month 6, Month 24, Month 60
  Level of fasting blood glucose
Incidence of untreated high blood pressure | Month 6, Month 24, Month 60
  Measure of systolic blood pressure
Incidence of hypertriglyceridemia | Month 6, Month 24, Month 60
  Level of triglyceridemia
Incidence of hyper-LDL-cholesterolemia | Month 6, Month 24, Month 60
  Level of LDL-cholesterolemia
Incidence of low level of physical activity | Month 6, Month 24, Month 60
  Questionnaire "Godin-Shephard Leisure-Time Physical Activity"
Incidence of insufficiency / deficiency of 25(OH) vitamin D (D2+D3) | Month 6, Month 24, Month 60
  Level of 25(OH) vitamin D (D2+D3)
Description of carcinogenic products consumption (tobacco, alcohol, cannabis) | Month 1, Month 6, Month 24, Month 60
  * Number of packages years
  * Questionnaire "DETA-Cage"
Evaluation of the Progression-free survival | Month 6, Month 24, Month 60
  Evaluation of the Progression-free survival
Evaluation of the Survival without an increase in the number of complications, among those studied | Month 6, Month 24, Month 60
  Evaluation of the Survival without an increase in the number of complications, among those studied
Evaluation of the event-free survival | Month 6, Month 24, Month 60
  Evaluation of the event-free survival
identification of demographiccs, clinical cancer, treatment-related parameters associated with complications occuring during follow-up | Month 1, Month 6, Month 24 and Month 60
  measurement of the association between demographics, clinical cancer and treatment-related parameters and the occurence of a type of complication during the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mauricette MICHALLET, PhD, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Leon Berard, Lyon, France

IPD SHARING:
Plan to Share IPD: No